CLINICAL TRIAL: NCT03693924
Title: A Retrospective Registry Study to Evaluate the Long-Term Efficacy and Safety of Superficial Radiation Therapy (SRT) for the Treatment of Recurrent Keloid Scars.
Brief Title: A Retrospective Evaluation of Superficial Radiation Therapy (SRT) and Keloid Scars.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sensus Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: SRTS-SRT-002
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Keloid Scar
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Radiation: SRT-100 — The SRT-100™ is a simple painless non-invasive in-office procedure that is approved by the U.S. Food and Drug Administration (U.S. FDA) to treat keloids caused by surgery or injury by delivering a precise, calibrated dose of Superficial Radiation Therapy (SRT) that only goes skin deep.

SUMMARY:
Keloid formation in response to skin trauma inflicts about 18 million individuals. A key impediment in successful treatment of keloids is that the predominant treatments, particularly surgical excision and shaving, tend to initiate the regrowth of the keloid at the excision site, and therefore, recurrence rates are high. There is much evidence to demonstrate that following surgical excision procedures with a course of radiation therapy can significantly reduce recurrence rates to as little as 10% or below. This retrospective study is to evaluate this claim.

DETAILED DESCRIPTION:
A keloid is an unsightly non-malignant tumor comprised of an abnormal proliferation of scar tissue that forms at the site of cutaneous injury (e.g. skin trauma such as cuts, abrasions and puncture wounds, burns or surgical incisions). It appears as a raised scar and does not regress and grows beyond the original margins of the scar. Keloids most commonly develop on the earlobes, neck, shoulders, chest, back, upper arms and cheeks. Keloids tends to grow slowly and continue to spread for weeks, months or even years. As a keloid grows, it may cause significant itching, pain, and tenderness upon touch, reduced mobility and emotional distress.

About 18 million people worldwide are genetically prone to form keloids in response to skin trauma, with equal gender distribution and greater susceptibility for darker-skinned individuals and those aged 10 to 30 years.

The greatest obstacle in treating keloids with many available surgical and non-surgical methods is that new keloids typically recur at the site of excision due to the treatment itself. For example, the recurrence rate using surgical excision alone is 45 to 100 percent.

Surgical excision followed by radiotherapy is a helpful treatment option for large and more difficult-to-treat keloids that cannot otherwise be treated by, or have failed, more conservative measures. It is thought that because keloid fibroblasts are sensitive to x-ray irradiation, it may prevent the recurrence of keloids by controlling fibroblast proliferation, arresting the cell cycle, and inducing premature cellular senescence. When surgical keloid excision is followed by Radiation Therapy, recurrence drops dramatically to 10% or below.

The SRT-100™ is a United States Food and Drug Administration (U.S. FDA) approved device for delivering a precise, calibrated dose of Superficial Radiation Therapy (SRT) to treat keloids caused by surgery or injury. This retrospective study has been designed to focus on efficacy and safety of the SRT-100™ for the treatment of recurrent keloid scars.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of keloid(s).
* Treatment with SRT-100™ of one or more keloids.
* At least 1 year since treatment end.
* Required retrospective data is existing and sufficient.

Exclusion Criteria

* Lesions of etiology other than keloids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients who were treated with the SRT-100™ for one or more recurrent keloids and who have at least 1 year of follow-up data.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-15 (Estimated); Primary Completion 2019-02-16 (Estimated); Study Completion 2019-02-16 (Estimated)

PRIMARY OUTCOMES:
Long-term recurrence rate | one year
  Recurrence rate will be calculated as the percentage of keloids that recurred at the treatment site following treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Berman, M.D., Principal Investigator